CLINICAL TRIAL: NCT06495853
Title: A Prospective Phase II Clinical Study on Continuous Circumferential Reinforcement of the Anastomotic Site With Laparoscopic Rectal Anastomosis to Prevent Complications.
Brief Title: Prospective Phase II Study on Continuous Circumferential Reinforcement of Laparoscopic Rectal Anastomosis to Prevent Complications
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ZHI-ZHONG PAN (Other)
Responsible Party: Sponsor-Investigator, ZHI-ZHONG PAN, Prof., Sun Yet-Sen University Cancer Center
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-FXY-182
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer; Anastomotic Leakage; Operation
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GroupA (Experimental): Patients with rectal cancer who did not receive neoadjuvant chemoradiotherapy and underwent rectal anterior resection with anastomotic reinforcement were included in Cohort A. The rectal cancer radical resection was performed in strict accordance with the principles of no-tumor technique and total mesorectal excision (TME) by experienced deputy chief physicians or higher from our research center. The procedure followed standard rectal cancer radical resection protocols. After rectal division using a linear stapler, an end-to-end anastomosis was performed using a circular stapler. For patients in the treatment group, anastomotic reinforcement was performed using absorbable Johnson & Johnson EB403 barbed sutures laparoscopically.Unless there were clear high-risk factors for anastomotic leakage preoperatively (e.g., diabetes, narrow pelvis, unsatisfactory anastomosis, positive colonic air leak test), ileostomy was not routinely performed in this group of patients.
  Interventions: Procedure: Continuous Circumferential Reinforcement of the Anastomotic
- Group B (Experimental): Patients who did not receive neoadjuvant chemoradiotherapy and underwent rectal anterior resection with anastomotic reinforcement were included in Cohort B. The rectal cancer radical resection was performed in strict accordance with the principles of no-tumor technique and total mesorectal excision (TME) by experienced deputy chief physicians or higher from our research center. The procedure followed standard rectal cancer radical resection protocols. After rectal division using a linear stapler, an end-to-end anastomosis was performed using a circular stapler. For patients in the treatment group, anastomotic reinforcement was performed using absorbable Johnson & Johnson EB403 barbed sutures laparoscopically.
  Since neoadjuvant chemoradiotherapy is a high-risk factor for postoperative anastomotic leakage, ileostomy was routinely performed in this group of patients to prevent severe intra-abdominal infections caused by anastomotic leakage.
  Interventions: Procedure: Continuous Circumferential Reinforcement of the Anastomotic

INTERVENTIONS:
Procedure: Continuous Circumferential Reinforcement of the Anastomotic — The reinforcement began on the right side of the anterior wall of the anastomosis, 0.5 cm from the anastomotic line, with continuous full-thickness sutures spaced 1 cm apart. The suture ended with fixation of the suture tail using non-absorbable vascular clips. The decision to perform splenic flexure mobilization depended on the anastomotic tension and the length of the resected bowel segment. The superior mesenteric artery and vein were divided at their roots.

SUMMARY:
Anastomotic leakage (AL) is one of the most severe complications following laparoscopic rectal cancer surgery. According to the International Study Group of Rectal Cancer (ISREC), AL is defined as a defect of intestinal wall integrity at the colorectal or coloanal anastomosis leading to a communication between the intra- and extraluminal compartments, including defects of the suture or staple lines of the neorectal reservoir. AL is classified into three grades based on clinical severity: Grade A, identified only radiologically without clinical symptoms; Grade B, presenting with localized or atypical peritonitis requiring antibiotics and local drainage but not surgery; and Grade C, causing severe peritonitis, systemic toxicity symptoms requiring urgent surgical intervention, and potentially leading to life-threatening situations.

AL can prolong hospitalization, necessitate reoperation, delay chemotherapy, increase local recurrence rates, and adversely affect survival and quality of life. Emergency surgical management of AL often requires meticulous peritoneal lavage and ileostomy, aiming for subsequent anastomotic healing or future digestive tract reconstruction. However, some patients face significant challenges due to postoperative adhesions and persistent anastomotic defects despite prolonged lavage.

Identified risk factors for AL after rectal cancer surgery include male gender, advanced age, hypertension, diabetes, smoking, and advanced TNM staging (III-IV). Additionally, preoperative chemoradiotherapy-induced bowel edema and fibrosis, bowel obstruction, and long-term malnutrition resulting in hypoproteinemia are significant contributors. Mechanical reinforcement of anastomoses using sutures or absorbable barbed sutures has been shown to significantly reduce AL rates in previous studies.

This single-center prospective phase II clinical trial aims to evaluate the efficacy and safety of continuous circumferential reinforcement using absorbable barbed sutures in laparoscopic rectal anastomosis to prevent AL. We will compare the incidence of AL and other postoperative complications between patients undergoing reinforced anastomosis and a control group receiving standard laparoscopic rectal anastomosis.

ELIGIBILITY:
Inclusion Criteria:

Histological Confirmation:

Diagnosed with rectal adenocarcinoma confirmed by histology.

Tumor Location:

MRI confirms a mid to upper rectal tumor, with the lower margin of the tumor located 6-12 cm from the anal verge.

Preoperative Staging:

Preoperative MRI staging indicates the presence or absence of MRF positivity and/or EMVI positivity; the surgical team assesses the tumor as resectable with an estimated R0 resection.

Bowel Obstruction:

No signs of bowel obstruction.

Neoadjuvant Chemoradiotherapy:

For patients who have received neoadjuvant chemoradiotherapy, complete radiotherapy and baseline imaging records must be available at this center.

Previous Treatments:

Surgical History:

No previous colorectal surgery.

Biological and Immunotherapy:

No prior treatment with biological drugs (e.g., monoclonal antibodies), immunotherapy (e.g., anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-PD-L2 antibodies, or anti-CTLA-4), or other investigational drugs.

Endocrine Therapy:

No restrictions on prior endocrine therapy.

Patient Characteristics:

Age:

Between 18 and 75 years old.

Performance Status:

ECOG performance status of 0-1 (see Appendix 3).

Life Expectancy:

Greater than 2 years.

Hematological Parameters:

WBC > 3×10^9/L; PLT > 80×10^9/L; Hb > 90 g/L.

Liver Function:

ALT and AST less than 2 times the upper limit of normal; bilirubin less than 1.5 times the upper limit of normal.

Renal Function:

Creatinine less than 1.5 times the upper limit of normal or creatinine clearance (CCr) ≥ 60 ml/min.

Exclusion Criteria:

Patients meeting any of the following conditions will be excluded from the study:

Need for Multiorgan Resection:

Patients requiring combined organ resection.

Preventive or Permanent Stoma:

Patients requiring preventive or permanent stoma.

Hartmann or Miles Procedures:

Patients requiring Hartmann's procedure or Miles' surgery.

Cardiac Conditions:

Arrhythmias requiring antiarrhythmic treatment (excluding β-blockers or digoxin), symptomatic coronary artery disease, localized myocardial ischemia (myocardial infarction within the last 6 months), or congestive heart failure beyond NYHA Class II.

Uncontrolled Hypertension:

Severe hypertension that is not well controlled by medication.

Infectious Diseases:

History of HIV infection or active chronic hepatitis B or C with high viral DNA copies.

Active Tuberculosis (TB):

Subjects with active pulmonary tuberculosis, currently undergoing anti-tuberculosis treatment, or having received anti-tuberculosis treatment within 1 year prior to screening.

Severe Infections:

Other active clinically severe infections (according to NCI-CTC version 5.0).

Evidence of Distant Metastasis:

Preoperative evidence of distant metastasis outside the pelvis.

Cachexia and Organ Failure:

Cachexia or decompensated organ function.

Radiotherapy History:

History of pelvic or abdominal radiotherapy.

Multiple Primary Colorectal Cancers:

Presence of multiple primary colorectal cancers.

Seizure Disorders:

Patients with seizures requiring treatment (e.g., steroids or antiepileptic therapy).

History of Other Malignancies:

History of other malignancies within the past 5 years, except for cured in situ cervical cancer or basal cell carcinoma of the skin.

Substance Abuse:

Substance abuse or medical, psychological, or social conditions that could interfere with the patient's participation in the study or the evaluation of study results.

Allergies:

Known or suspected allergies to the investigational drug or any drug related to the study.

Unstable Conditions:

Any unstable condition or situation that might jeopardize patient safety and compliance.

Pregnancy or Lactation:

Women who are pregnant or breastfeeding, and women of childbearing potential not using adequate contraceptive measures.

Informed Consent:

Refusal to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Clinically and Radiologically Confirmed Anastomotic Leakage within 30 Days Postoperatively | 30-days after surgery
  Clinical and radiological assessment of anastomotic leakage within 30 days postoperatively, including Grade A and B leaks detected through imaging without clinical symptoms, as well as Grade C leaks with clear clinical manifestations.

SECONDARY OUTCOMES:
Time to First Postoperative Flatus | 3-days after surgery
  Time to First Postoperative Flatus
Time to First Postoperative Oral Intake | 3-days after surgery
  This refers to the duration from the end of surgery until the patient is able to tolerate oral intake of food or liquids.
Incidence of Postoperative Intra-abdominal Hemorrhage | 14-days after surgery
  This refers to the frequency at which patients experience bleeding within the abdominal cavity following surgery. It is typically assessed through clinical signs, imaging studies, and the need for interventions such as transfusions or reoperations.
Incidence of Postoperative Anastomotic Hemorrhage | 14-days after surgery
  This refers to the frequency at which patients experience bleeding at the site of the anastomosis following surgery. It is typically evaluated based on clinical symptoms, endoscopic findings, or imaging studies, and may require interventions such as endoscopic hemostasis, transfusions, or reoperation.
Incidence of Postoperative Anastomotic Stricture | 60-days after surgery
  This refers to the frequency at which patients develop a narrowing at the anastomotic site following surgery. This condition can be identified through symptoms such as difficulty in passing stool, abdominal pain, or diagnosed via endoscopy or imaging studies. It may require interventions such as balloon dilation, stenting, or surgical revision.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorectal Department,SunYat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No